## COVID-19 Booster Readiness Survey (NCT05529030)

Statistical Analysis Plan

September 6, 2022

## **Statistical Analysis Plan**

As of the writing of this plan, the survey has been distributed, but the data have not been examined.

Since the findings of this administrative survey are immediately needed for hospital operations, the researchers will examine the data and conduct descriptive analyses (e.g., number of people interested in a bivalent booster broken down by categories like job role; reasons for hesitancy) as early as 5 days after the start of the survey (September 6).

Randomized data will not be examined other than checking that the random assignment yielded groups of similar size. There are 4 randomly assigned groups:

- V1: Standard question
- V2: Question with salient Omicron message
- V3: Question with patient protection message (patient-facing participants only)
- V4: Question with salient Omicron message and patient protection message (patient-facing participants only)

The primary analysis of the primary outcome (effect of experimental group on interest in a bivalent booster; yes/no/unsure) will not be conducted until 14 days after the start of the survey (September 15). The extended study period will allow as much data to be collected as is reasonable, even if the deadline of the survey has passed (September 9).